CLINICAL TRIAL: NCT00376285
Title: A Phase 1, Randomized, Investigator and Subject Blind, Sponsor Open Study to Determine the Effects of Fenofibrate on the Safety, Toleration and Efficacy Biomarkers of CP-742,033 When Co-Administered in Otherwise Healthy Obese Adult Subjects
Brief Title: Effects of Fenofibrate on the Safety, Toleration and Efficacy Biomarkers of CP-742,033
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A5431015
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Fenofibrate

INTERVENTIONS:
Drug: CP-742,033
Drug: Fenofibrate

SUMMARY:
The purpose of this study is to determine whether fenofibrate effects the toleration, safety, or efficacy biomarkers of CP-742,033, a drug being developed for the treatment of obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 30-40 kg/m2

Exclusion Criteria:

* Women of childbearing potential

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-11

PRIMARY OUTCOMES:
Toleration and safety

SECONDARY OUTCOMES:
Efficacy biomarkers, serum lipids

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5431015&StudyName=Effects+of+Fenofibrate+on+the+Safety%2C+Toleration+and+Efficacy+Biomarkers+of+CP%2D742%2C033